CLINICAL TRIAL: NCT03412786
Title: A Phase I Study of the Bcl-XL_42-CAF09b Vaccine to Test Safety and Immunological Effect in Patients With Prostate Cancer With Lymph Node Metastases
Brief Title: Bcl-XL_42-CAF09b Vaccination for Patients With Prostate Cancer With Lymph Node Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Inge Marie Svane, Prof., MD, Herlev Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UR1534
Record Dates: First submitted 2018-01-02; First posted 2018-01-26 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Masking Description: Not a randomized study. The first 10 patients included will be treated in arm A - the last 10 will be treated in arm B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: IM followed by IP (Experimental): Will be administered first 3 vaccines biweekly IM and thereafter 3 vaccines biweekly IP.
  Interventions: Biological: Bcl-Xl_42-CAF09b vaccine
- Arm B: IP followed by IM (Experimental): Will be administered first 3 vaccines biweekly IP and thereafter 3 vaccines biweekly IM.
  Interventions: Biological: Bcl-Xl_42-CAF09b vaccine

INTERVENTIONS:
Biological: Bcl-Xl_42-CAF09b vaccine — The vaccine consists of 0.05 mg peptide (bcl-xl_42) and 625 μg DDA, 125 μg MMG og 31 μg Poly I:C (CAF09b) mixed in a 0.5 ml emulsion

SUMMARY:
In this Phase I study, patients with hormone-sensitive Prostate Cancer (PC) and lymph node metastases are treated with the cancer vaccine Bcl-xl_42-CAF09b. The aim of the study is to clarify the safety and toxicity of the vaccine and also the immunological effect.

The vaccine Bcl-xl_42-CAF09b is composed of the peptide Bcl-xl_42 and the adjuvant CAF09b. The B-cell lymphoma extra large protein (Bcl-xl) protein plays a vital role in the cancer cell's ability to avoid programmed cell death (apoptosis) and is upregulated in a variety of cancerous diseases. Bcl-xl_42 is a peptide fragment of the full protein and preclinical studies have shown that vaccination with this peptide (Bcl-xl) can activate the immune system and thereby lead to the death of cancer cells. In order to improve the activation of the immune system, adjuvant CAF09b is added; Preclinical studies have shown that special intraperitoneal (IP) injections of CAF09b improve the activation of the immune system.

DETAILED DESCRIPTION:
Background:

In this Phase I study, patients with hormone-sensitive Prostate Cancer (PC) and lymph node metastases are treated with the cancer vaccine Bcl-xl_42-CAF09b. The aim of the study is to clarify the safety and toxicity of the vaccine and also the immunological effect.

Patients included should be on Bicalutamid treatment upon inclusion. The vaccine Bcl-xl_42-CAF09b is composed of the peptide Bcl-xl_42 and the adjuvant CAF09b. The B-cell lymphoma extra large protein (Bcl-xl) protein plays a vital role in the cancer cell's ability to avoid programmed cell death (apoptosis) and is upregulated in a variety of cancerous diseases. Bcl-xl_42 is a peptide fragment of the full protein and preclinical studies have shown that vaccination with this peptide (Bcl-xl) can activate the immune system and thereby lead to the death of cancer cells.

In order to improve the activation of the immune system, adjuvant CAF09b is added; Preclinical studies have shown that special intraperitoneal (IP) injections of CAF09b improve the activation of the immune system.

The CAF09 adjuvant has been developed by Statens Serum Institut (SSI). It is a three-component adjuvant system, composed of cationic liposomes (DDA-MMG1) with complex bound synthetic double-stranded RNA (Poly(I:C)2). The adjuvant was developed as a means to induce cytotoxic CD8+ T-cell responses against vaccine antigens and intended for use in vaccines against disease targets such as cancers, human immunodeficiency virus or Hepatitis C virus. The Poly(I:C) component has previously been in clinical studies as a cancer treatment. Poly(I:C) is known for its pyrogenic activity but upon formulation in the cationic liposome system, CAF09, the pyrogenic effect is significantly reduced.

Methods:

20 patients will be included in this phase I trial. 10 patients will be included in arm A and 10 patients in arm B. Arm a will recieve 3 vaccines every second week IM and thereafter 3 vaccines every second week IP. Arm B will first receive 3 vaccines every second week IP and thereafter every second week IM. All 20 patients will recieve 6 vaccines all in all. This is not randomized - the first 10 patients included will be in arm A and the last 10 patients included will be in arm B.

Patients will be followed with clinical controls every second week.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically Verified Adenocarcinoma Prostatae
3. Diagnostic and / or histologically verified lymph node metastases
4. ECOG Performance Status ≤2
5. Primary anti-androgen treatment started
6. Adequate haematological, renal and hepatic function:

   1. Neutrophil granulocytes ≥ 1.5 x 109 / l
   2. Platelet counts ≥ 100 x 109 / l
   3. hemoglobin ≥ 5.6 mmol / l
   4. Serum creatinine ≤ 1.5 times upper normal limit
   5. AST or ALAT ≤ 2.5 times upper normal limit
   6. serum bilirubin ≤ 1.5 times upper normal limit
   7. Alkaline phosphatase ≤ 2.5 times upper normal limit
   8. INR <1.5 / PP <40

Exclusion Criteria:

1. Verified bone or visceral metastases
2. Serious allergy or previous anaphylactic reactions
3. Known hypersensitivity to any of the active substances or to any of the excipients.
4. Other malignant disease within the last three years, rendering planocellular and basocellular skin carcinoma
5. Known infection with HIV, hepatitis B and C virus, regardless of whether the infection is kept calm with medical treatment
6. Severe medical disorder, severe asthma, severe COPD, poorly regulated cardiovascular disease or diabetes
7. Active autoimmune disease, e.g. autoimmune neutropenia / thrombocytopenia or hemolytic anemia, systemic lupus erythematosus, scleroderma, myasthenia gravis, goodpasture syndrome, Addison's disease, Hashimoto's thyroiditis, active grave disease, morbus chrohn or ulcerative colitis
8. Major gastrointestinal surgical procedures within the last 3 months
9. Previous treatment with other cancer vaccine
10. Concomitant immunosuppressive treatment including prednisolone and methotrexate
11. Ongoing anticoagulant treatment (treatment with acetylsalicylic acid and clopidogrel is allowed)
12. Psychiatric disease which, according to the investigator's discretion, may affect compliance
13. Co-administration with other experimental drugs.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Number and type of reported adverse events | 0-30 weeks
  Determine the safety of the Bcl-XL_42-CAF09b vaccine for patients with prostate cancer with lymph node involvement who are on Bicalutamid treatment by reporting adverse events according to CTCAE v. 4.0

SECONDARY OUTCOMES:
Treatment related immune responses | Up to 24 months
  To evaluate the immunological impact of the treatment in both arm A and arm B. Elispot and tetramer staining methods will be Applied to identify Bcl-XL_42 peptide specific T cells in the blood over time

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie svane, Study Director — Sponsor GmbH
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mork SK, Kongsted P, Westergaard MCW, Albieri B, Granhoj JS, Donia M, Martinenaite E, Holmstrom MO, Madsen K, Kverneland AH, Kjeldsen JW, Holmstroem RB, Lorentzen CL, Norgaard N, Andreasen LV, Wood GK, Christensen D, Klausen MS, Hadrup SR, Thor Straten P, Andersen MH, Svane IM. First in man study: Bcl-Xl_42-CAF(R)09b vaccines in patients with locally advanced prostate cancer. Front Immunol. 2023 Mar 14;14:1122977. doi: 10.3389/fimmu.2023.1122977. eCollection 2023. PMID 36999039